CLINICAL TRIAL: NCT02979717
Title: The Effect of a High Protein, High Fibre Shake Pre-load on Measures of Satiety and Subsequent Energy Intake in Healthy Overweight and Obese Subjects: An Acute Randomized, Crossover, Double-blind Placebo-controlled Study
Brief Title: The Effect of a High Protein, High Fibre Shake Pre-load on Measures of Satiety and Subsequent Energy Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beachbody (Industry)
Collaborators: Glycemic Index Laboratories, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: GIL-1653
Record Dates: First submitted 2016-11-28; First posted 2016-12-02 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Overweight and Obesity
Keywords: satiety; protein; fiber
MeSH Terms: conditions — Overweight; Obesity | interventions — Diet, Protein-Restricted

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- high protein, high fiber (Experimental): Participants receive a high protein, high fiber dietary supplement pre-load
  Interventions: Dietary Supplement: High protein, high fiber dietary supplement
- Low protein, low fiber (Placebo Comparator): Participants receive a low protein, low fiber isocaloric pre-load
  Interventions: Other: Low protein, low fiber comparator

INTERVENTIONS:
Dietary Supplement: High protein, high fiber dietary supplement
  Arms: high protein, high fiber
Other: Low protein, low fiber comparator
  Arms: Low protein, low fiber

SUMMARY:
The objective of this study is to determine the effect of a high protein, high fiber supplement pre-load on energy intake at a subsequent meal compared to a low fiber, high carbohydrate Control product in healthy overweight and obese subjects. The investigators hypothesize the high protein, high fiber pre-load will result in reduced energy intake at a subsequent meal compared to low protein, low fiber.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant, non-lactating females, 18-50 years of age, inclusive
2. Body mass index (BMI) between 27 and 33 kg/m² inclusive at screening.
3. Blood pressure < 130/85.
4. Willing to maintain habitual diet, physical activity pattern, and body weight throughout the trial.
5. Willing to abstain from strenuous exercise, consumption of alcoholic drinks and caffeine-containing food/drinks 24 hours before study days and during study days (until study completion for that day).
6. Willing to maintain current dietary supplement (if applicable) use throughout the trial. On test days, subject agrees not to take any dietary supplements until dismissal from the GI labs. Failure to comply will result in a rescheduled test visit.
7. Absence of health conditions that would prevent fulfillment of study requirements as judged by the Investigator on the basis of medical history.
8. Understanding the study procedures and willing to provide informed consent to participate in the study and authorization to release relevant protected health information to the study investigator.
9. Female subjects are willing to use a contraceptive method to avoid pregnancy during the study period.

Exclusion Criteria:

1. Failure to meet any one of the inclusion criteria
2. Smokers
3. Known history of AIDS, hepatitis, a history or presence of clinically important endocrine (including Type 1 or Type 2 diabetes mellitus), cardiovascular (including, but not limited to, atherosclerotic disease, history of myocardial infarction, peripheral arterial disease, stroke), pulmonary, biliary or GI disorders.
4. Use of medications known to influence carbohydrate metabolism, gastrointestinal function or appetite, including, but not limited to adrenergic blockers, blood thinners, diuretics, thiazolidinediones, metformin, antibiotics and systemic corticosteroids within 4 weeks of the screening visit, or with any condition which might, in the opinion of Dr. Wolever, the president of GI labs, either: 1) make participation dangerous to the subject or to others, or 2) affect the results.
5. Major trauma or surgical event within 3 months of screening.
6. Unwillingness or inability to comply with the experimental procedures and to follow GI Labs safety guidelines.
7. Known intolerance, sensitivity or allergy to any ingredients in the study products.
8. Extreme dietary habits, as judged by the Investigator (i.e. Atkins diet, very high protein diets, etc)..
9. Change in body weight of >3.5kg within 4 weeks of the screening visit.
10. Presence of any signs or symptoms of an active infection within 5 d prior to any test visit. If an infection occurs during the study period, test visits should be rescheduled until all signs and symptoms have resolved and any treatment (i.e. antibiotic therapy) has been completed at least 5 d prior to each test visit.
11. History of cancer in the prior two years, except for non-melanoma skin cancer.
12. Exposure to any non-registered drug product within 30 d prior to screening.
13. Pregnancy or breastfeeding
14. Any history of an eating disorder (e.g., anorexia nervosa, bulimia nervosa, binge eating) diagnosed by a health professional

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2016-11-23 (Actual); Primary Completion 2017-03-14 (Actual); Study Completion 2017-03-14 (Actual)

PRIMARY OUTCOMES:
Energy intake (total kilocalories) at meal subsequent to intervention pre-load | 1 hour post-intervention
  Participants will consume an ad-libitum pizza meal for 30 minutes, 30 minutes following ingestion of the pre-load intervention. At the end of the 30 minute pizza meal, total caloric intake will be recorded.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) Appetite Questionnaire on scale of 0-100 | pre-intervention; 10, 20, 30, 60 min post-intervention
  A standard VAS Appetite questionnaire will be completed by subjects before pre-load intervention, and at indicated time intervals. The 4 questions assess hunger, fullness, desire to eat, and prospective consumption. Each of the questions on the VAS is a 100 mm line anchored at each end with opposing statements. Participants mark a vertical line on the line at a point that they felt reflect their feelings at the moment the test was taken. Scores will be assessed by measuring the distance between the intersection of the vertical line with the line and the left end of the line.
Visual Analog Scale (VAS) Cravings Questionnaire on scale of 0-100 | pre-intervention; 10, 20, 30, 60 min post-intervention
  A standard VAS Cravings questionnaire will be completed by subjects before pre-load intervention, and at indicated time intervals. The 4 questions assess cravings for sweet, salty, savory, and fatty. Each of the questions on the VAS is a 100 mm line anchored at each end with opposing statements. Participants mark a vertical line on the line at a point that they felt reflect their feelings at the moment the test was taken. Scores will be assessed by measuring the distance between the intersection of the vertical line with the line and the left end of the line.
Subjective Physical Comfort Questionnaire on scale of 0-100 | pre-intervention; immediately post-intervention; 30 min post-intervention
  This questionnaire assesses Gastrointestinal symptoms including Bloating, Belching, Nausea, Diarrhea, and Flatulence. Participants identify if they are currently experiencing the symptom (Yes/No) and if yes, rate the severity of the symptom (Low to High) on a 100 mm scale (0-100). Measures will be made from the left side of the scale, similar to Appetite and Cravings questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Wolever, PhD,DM(Oxon), Principal Investigator — Glycemic Index Laboratories, Inc
Locations (1):
- Glycemic Index Laboratories, Inc., Toronto, Ontario, Canada

REFERENCES:
- [Derived] Sharafi M, Alamdari N, Wilson M, Leidy HJ, Glynn EL. Effect of a High-Protein, High-Fiber Beverage Preload on Subjective Appetite Ratings and Subsequent Ad Libitum Energy Intake in Overweight Men and Women: A Randomized, Double-Blind Placebo-Controlled, Crossover Study. Curr Dev Nutr. 2018 Jun 23;2(6):nzy022. doi: 10.1093/cdn/nzy022. eCollection 2018 Jun. PMID 29955731